CLINICAL TRIAL: NCT04722042
Title: Place-based Mapping in Electric-acoustic Stimulation Listeners
Brief Title: Place-based Mapping in EAS Listeners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-3022; R21DC018389 (NIH)
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-07

CONDITIONS: Cochlear Implant

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and testing audiologist were blinded to the randomized map for Arm 1 (cochlear implant users with default maps) and Arm 2 (cochlear implant users with place-based maps). Arm 3 is normal hearing participants listening to simulations of default and place-based maps.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cochlear implant participants with Default maps (Other): The default frequency filters assigned by the clinical software
  Interventions: Other: default mapping
- Cochlear implant participants with Place-Based maps (Experimental): Frequency filters adjusted to align with the cochlear place frequency
  Interventions: Other: place-based mapping
- Normal hearing controls listening to simulations (Other): Normal hearing controls listening to simulations of default and place-based maps.
  Interventions: Other: place-based mapping; Other: default mapping

INTERVENTIONS:
Other: place-based mapping — Adjusting the electric frequency filters to align with the cochlear place frequency
  Arms: Cochlear implant participants with Place-Based maps; Normal hearing controls listening to simulations
Other: default mapping — Default frequency filter assignments
  Arms: Cochlear implant participants with Default maps; Normal hearing controls listening to simulations

SUMMARY:
Purpose: Investigate monaural and binaural hearing in electric-acoustic stimulation (EAS) users with place-based versus default maps.

Participants: Cochlear implant recipients and normal-hearing listeners Procedures (methods): This is a prospective, longitudinal investigation of the monaural and binaural outcomes (such as speech perception, spatial hearing, and/or subjective benefit) of cochlear implant recipients listening with different programs. The programs will incorporate different patient and device variables to determine the effect on cochlear implant recipient outcomes.

ELIGIBILITY:
Cochlear implant participants

Inclusion Criteria:

* 18-80 years of age at implantation, identify English as native language, Medical Electronics (MED-EL) array recipient, and a postoperative unaided detection threshold of less than or equal to 65 decibel (dB) hearing level (HL) at 125 Hz

Exclusion Criteria:

* Report or present with a cognitive delay or impairment

Normal-hearing controls

Inclusion Criteria:

* 18-80 years of age at time of testing, unaided detection thresholds of 35 dB HL or better from 500-4000 Hz, identify English as native language

Exclusion Criteria:

* Report or present with a cognitive delay or impairment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret T Dillon, AuD, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Kevin D Brown, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC ENT at Carolina Crossing, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: beginning 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Result] Dillon MT, Canfarotta MW, Buss E, Rooth MA, Richter ME, Overton AB, Roth NE, Dillon SM, Raymond JH, Young A, Pearson AC, Davis AG, Dedmon MM, Brown KD, O'Connell BP. Influence of Electric Frequency-to-Place Mismatches on the Early Speech Recognition Outcomes for Electric-Acoustic Stimulation Users. Am J Audiol. 2023 Mar;32(1):251-260. doi: 10.1044/2022_AJA-21-00254. Epub 2023 Feb 17. PMID 36800505
- [Result] Dillon MT, O'Connell BP, Canfarotta MW, Buss E, Hopfinger J. Effect of Place-Based Versus Default Mapping Procedures on Masked Speech Recognition: Simulations of Cochlear Implant Alone and Electric-Acoustic Stimulation. Am J Audiol. 2022 Jun 2;31(2):322-337. doi: 10.1044/2022_AJA-21-00123. Epub 2022 Apr 8. PMID 35394798
- [Result] Dillon MT, Canfarotta MW, Buss E, Hopfinger J, O'Connell BP. Effectiveness of Place-based Mapping in Electric-Acoustic Stimulation Devices. Otol Neurotol. 2021 Jan;42(1):197-202. doi: 10.1097/MAO.0000000000002965. PMID 33885267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three study arms: 1) Participants with a cochlear implant randomized to listen with a default map (Arm 1), 2) Participants with a cochlear implant randomized to listen with a place-based map, and 3) Participants with normal hearing who listened to simulations of both maps (control group).
Pre-assignment Details: Participants with cochlear implants were randomized to one of two groups (arms): Arm 1 (default maps) or Arm 2 (place-based maps)
  Participants with normal hearing (Arm 3; control group) listened to simulations of default and place-based maps.
Groups:
- Default: The default frequency filters assigned by the clinical software
  default mapping: Default frequency filter assignments
- Place-based: Frequency filters adjusted to align with the cochlear place frequency
  place-based mapping: Adjusting the electric frequency filters to align with the cochlear place frequency
- Normal Hearing Control: age-matched listeners with normal hearing in both ears
Period: Overall Study
Arm/Group | Default | Place-based | Normal Hearing Control
Started | 13 | 11 | 15
Completed | 11 | 10 | 15
Not Completed | 2 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Normal Hearing Control Group: age-matched listeners with normal hearing in both ears
- Total: Total of all reporting groups
Arm/Group | Default | Place-based | Normal Hearing Control Group | Total
Number analyzed (Participants) | 13 | 11 | 15 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 7 | 5 | 11 | 23
  >=65 years | 6 | 5 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (14) | 58 (17) | 54 (16) | 60 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 11 | 25
  Male | 5 | 5 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 15 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 5
  White | 13 | 7 | 13 | 33
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 11 | 15 | 39
Unaided Threshold at 125 Hz [Mean (Standard Deviation); unit: decibels] | 38 (12) | 30 (13) | 15 (7) | 34 (13)

OUTCOME MEASURES:

1. Primary Outcome: Monaural Perception for Participants With Cochlear Implants (Arms 1 and 2) Over Time
Description: Monaural perception (e.g., word recognition in quiet) will be assessed at defined intervals (e.g., activation, and 1, 3, 6, and 12 months post-activation). Performance (e.g., percent correct) will be compared within-subject and between group over the study intervals.
  This procedure is specific to Arm 1 (participants with default maps) and Arm 2 (participants with place-based maps).
Time Frame: Up to 12 months post-activation
Population: This procedure is specific to Arm 1 (participants with default maps) and Arm 2 (participants with place-based maps).
Measure: Mean (Standard Deviation); unit: percent of words correctly repeated
Arm/Group | Default | Place-based
Number analyzed (Participants) | 11 | 10
percent of words correctly repeated
  activation | 18 (16) | 10 (14)
  1 month | 40 (23) | 34 (22)
  3 months | 49 (20) | 45 (16)
  6 months | 53 (22) | 50 (19)
  12 months | 56 (26) | 54 (15)
Statistical Analysis 1: Comparison: Default vs Place-based; comparison of word recognition over time (activation, and 1, 3, 6, and 12 months post-activation) between groups (default versus place-based); Test type: Superiority; p = 0.557, ANOVA

2. Primary Outcome: Binaural Hearing Abilities Over Time (Noise to the Study Ear Minus Noise From the Front)
Description: Binaural hearing abilities (e.g., spatial release from masking) will be assessed at defined intervals (e.g., 1, 3, 6, and 12 months post-activation). Performance (e.g., percent correct) will be compared within-subject and between group over the study intervals.
  This procedure is specific to Arm 1 (participants with default maps) and Arm 2 (participants with place-based maps).
Time Frame: Up to 12 months post-activation
Population: This procedure is specific to Arm 1 (participants with default maps) and Arm 2 (participants with place-based maps).
Measure: Mean (Standard Deviation); unit: percent of words correctly repeated
Arm/Group | Default | Place-based
Number analyzed (Participants) | 11 | 10
percent of words correctly repeated
  1 month | 10 (21) | 19 (23)
  3 month | 20 (19) | 24 (17)
  6 month | 10 (19) | 20 (24)
  12 month | 18 (21) | 28 (14)
Statistical Analysis 1: Comparison: Default vs Place-based; comparison of spatial release from masking over time (1, 3, 6, and 12 months post-activation) between the groups (default versus place-based); Test type: Superiority; p = 0.208, ANOVA

3. Primary Outcome: Binaural Hearing Abilities Over Time (Noise to the Non-study Ear Minus Noise From the Front)
Description: as for outcome 2
Time Frame: Up to 12 months post-activation
Population: This procedure is specific to Arm 1 (participants with default maps) and Arm 2 (participants with place-based maps).
Measure: Mean (Standard Deviation); unit: percent of words correctly repeated
Arm/Group | Default | Place-based
Number analyzed (Participants) | 11 | 10
percent of words correctly repeated
  1 month | 6 (14) | 0 (11)
  3 month | 15 (11) | 10 (14)
  6 month | 14 (14) | 5 (14)
  12 month | 16 (16) | 17 (18)
Statistical Analysis 1: Comparison: Default vs Place-based; comparison of spatial release from masking between the groups over time; Test type: Superiority; p = 0.126, ANOVA

4. Secondary Outcome: Perceived Abilities Over Time
Description: Perceived abilities will be assessed with questionnaires (e.g., Speech, Spatial, and Qualities of hearing scale; SSQ) at defined intervals (e.g., activation, and 1, 3, 6, and 12 months post-activation). A subject indicates his/her perceived abilities for each question on the SSQ using a Likert scale, with a range of 0-10 (with 10 indicating better perceived abilities). Responses will be compared between group over the study intervals.
  This procedure is specific to Arm 1 (participants with default maps) and Arm 2 (participants with place-based maps).
Time Frame: Up to 12 months post-activation
Population: This procedure is specific to Arm 1 (participants with default maps) and Arm 2 (participants with place-based maps).
  One participant in the place-based group did not complete the SSQ questionnaire at the 6 month post-activation visit.
Measure: Mean (Standard Deviation); unit: score on scale of 1 (worst) to 10 (best)
Arm/Group | Default | Place-based
Number analyzed (Participants) | 11 | 10
score on scale of 1 (worst) to 10 (best)
  preop | 4 (1) | 4 (1)
  1 month | 5 (2) | 5 (2)
  3 months | 5 (2) | 6 (2)
  6 months: number analyzed (Participants) | 11 | 9
  6 months | 5 (2) | 6 (2)
  12 months | 6 (2) | 7 (1)
Statistical Analysis 1: Comparison: Default vs Place-based; comparison of perceived benefit between the groups over time; Test type: Superiority; p = 0.369, ANOVA

5. Other Pre Specified Outcome: Word Recognition With Default Versus Place-based Maps for Participants With Normal Hearing
Description: Participants with normal hearing (Arm 3) listening to simulations of default versus place-based maps.
  All procedures completed at baseline (one visit that was ~ 20 minutes in duration). There were no follow-up visits.
Time Frame: All procedures completed at baseline (one visit that was ~ 20 minutes in duration).
Population: Arm 3: Participants with normal hearing listening to simulations of default versus place-based maps One participant did not complete this task
Measure: Mean (Standard Error); unit: percent of words correctly repeated
Groups:
- Normal Hearing Control: normal hearing controls
Arm/Group | Normal Hearing Control
Number analyzed (Participants) | 14
percent of words correctly repeated
  default map | 64 (28)
  place-based map | 78 (23)
Statistical Analysis 1: Comparison: Normal Hearing Control; Test type: Superiority; p = 0.006, t-test, 2 sided

6. Other Pre Specified Outcome: Vowel Recognition for Participants With Normal Hearing
Description: Vowel recognition for participants with normal hearing controls listening to simulations of default versus place-based maps.
  All procedures completed at baseline (one visit that was ~ 20 minutes in duration). There were no additional visits.
Time Frame: All procedures completed at baseline (one visit that was ~ 20 minutes in duration).
Population: Arm 3: Participants with normal hearing listening to simulations of default versus place-based maps
Measure: Mean (Standard Deviation); unit: percent of vowels correctly repeated
Arm/Group | Normal Hearing Control
Number analyzed (Participants) | 15
percent of vowels correctly repeated
  default map | 49 (17)
  place-based map | 60 (13)
Statistical Analysis 1: Comparison: Normal Hearing Control; Test type: Superiority; p < 0.001, t-test, 2 sided

7. Other Pre Specified Outcome: Sentence Understanding in Noise for Participants With Normal Hearing
Description: Sentence understanding in noise for participants with normal hearing controls listening to simulations of default versus place-based maps
  All procedures completed at baseline (one visit that was ~ 20 minutes in duration). There were no additional visits.
Time Frame: All procedures completed at baseline (one visit that was ~ 20 minutes in duration).
Population: Arm 3: Participants with normal hearing listening to simulations of default versus place-based maps
Measure: Mean (Standard Deviation); unit: percent of words correctly repeated
Arm/Group | Normal Hearing Control
Number analyzed (Participants) | 15
percent of words correctly repeated
  default map | 52 (24)
  place-based map | 63 (18)
Statistical Analysis 1: Comparison: Normal Hearing Control; Test type: Superiority; p = 0.02, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 year from cochlear implant activation for participants in Arms 1 and 2. Participants in Arms 1 and 2 were cochlear implant recipients who were followed for 1 year after cochlear implant activation. Single visit (baseline) for participants in Arm 3. Participants in Arm 3 had normal hearing and listened to simulations of default and place-based maps during one visit.
Groups:
- Cochlear Implant Users With Default Maps: The default frequency filters assigned by the clinical software
  default mapping: Default frequency filter assignments
- Cochlear Implant Users With Place-based Maps: Frequency filters adjusted to align with the cochlear place frequency
  place-based mapping: Adjusting the electric frequency filters to align with the cochlear place frequency
- Normal Hearing Controls: Normal hearing participants listening to simulations of default and place-based maps.
Arm/Group | Cochlear Implant Users With Default Maps | Cochlear Implant Users With Place-based Maps | Normal Hearing Controls
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-02-17): https://cdn.clinicaltrials.gov/large-docs/42/NCT04722042/Prot_SAP_001.pdf
  • Informed Consent Form (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT04722042/ICF_000.pdf